CLINICAL TRIAL: NCT04036370
Title: The Effect of Continuous Pectoral Nerve Block on Postoperative Analgesia Consumption in Breast Cancer Surgery
Brief Title: Continuous Pectoral Nerve Block in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Arzu Karaveli, University of Health Sciences Antalya Training and Research Hospital, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13/21
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-07

CONDITIONS: Nerve Blocks; Breast Surgery; Postoperative Pain
Keywords: pectoral nerve block (pecs block); breast cancer; postoperative pain; numeric rating scale score (NRS score)
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomised Controlled
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS group (Active Comparator): In addition to routine analgesic protocol; before anaesthesia induction; following the PECS I + II block, a continuous infusion catheter will be placed at the PECS II block level under the guidance of USG, and local anesthetic infusion will be started via the catheter at the end of the operation.
  Interventions: Procedure: PECS group
- Control group (Sham Comparator): Peroperative and postoperative routine analgesic protocol will be performed with no additional intervention (block).
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: PECS group — Pecs block performed using ultrasound guidance. Standard pain follow up and monitorization will be performed.
  Arms: PECS group
Other: Control group — Standard pain follow up and monitorization will be performed.
  Arms: Control group

SUMMARY:
The purpose of the study is to evaluate the effect of continuous pectoral nerve block on postoperative analgesia consumption in breast cancer surgery.

DETAILED DESCRIPTION:
Pectoral nerve block has been developed as an alternative to thoracic paravertebral and/or thoracic epidural blocks in recent years. It is frequently applied for postoperative analgesia in breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I-II
* 18-65 years
* Body mass index (BMI) ≤40 kg/m2
* Elective breast cancer surgery

Exclusion Criteria:

* ASA ≥4
* under 18 years of age or over 65 years of age
* declining to give written informed consent
* history of allergy to the local anesthetics
* contraendications of peripheral block or local anesthetic infiltration (local infection, coagulopathy, etc)
* history of breast surgery
* treatment due to psychiatric disorder
* history of treatment for chronic pain
* history of nerve blocks in order to treat postoperative pain

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
analgesia consumption | 12 hours
  postoperative 12 hours

SECONDARY OUTCOMES:
analgesia consumption | during the surgery
  intraoperative
postoperative Numeric Rating Scale (NRS) score | 0, 1, 3, 6, 9, 12 hours
  postoperative pain assessment will be performed using NRS score (NRS 0=no pain, NRS 10= most severe possible). The NRS scores will be recorded at postoperative 0, 1, 3, 6, 9, 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Antalya TRH
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Blanco R, Parras Maldonado T. Reply to the article entitled "Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery". Reply of the authors. Rev Esp Anestesiol Reanim. 2013 May;60(5):296-7. doi: 10.1016/j.redar.2013.01.002. Epub 2013 Feb 27. No abstract available. PMID 23453236
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971